CLINICAL TRIAL: NCT03234205
Title: Measurements of Myocardial Relaxation Time by MRI During Respiration
Acronym: ARTEMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2011-A00154-37
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: Heart Transplantation
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI scan during free respiration (Experimental)
  Interventions: Device: MRI scan

INTERVENTIONS:
Device: MRI scan — MRI standard protocol with addition of:
  * a second clinical respiratory belt besides belt usually installed for clinical examination
  * a second clinical electrocardiogram sensor besides sensor usually installed for clinical examination
  * 12 sequences during free respiration are added lasting supplementary 15 minutes
  * Use of cardiac antennae usually used for cardiac MRI scans

SUMMARY:
Measurement of T2 transversal relaxation time by magnetic resonance has a major interest in cardiac imagery. It has been initially used for quantitative evaluation of heart viability and more recently for edema characterization. It allows to prematurely detect a cardiac transplant rejection. This technique needs successively around ten FSE sequences during apnea. Weak reproducibility of successive apneas and discomfort of patient limit the precision of this measurement and consequently its use in standard care. The ARTEMIS study method allows the examination during free respiration without prolonging the duration of examination compared to the examination during apnea. Moreover, image processing is simplified and correction of respiratory movements renders results more reliable.

This is a pilot study of evaluation of ARTEMIS technique of image reconstruction. ARTEMIS is a method of MRI image reconstruction for measurements of T2 transversal relaxation. It allows to obtain diagnostic images without movement artifacts.

The primary objective si to show the feasibility of ARTEMIS method for measurement of myocardial T2 relaxation time during free respiration in cardiac transplant patients.

The secondary objective is to collect quantitative data to compare ARTEMIS method of measurement of T2 during free respiration and standard clinical practice during apnea.

ELIGIBILITY:
Inclusion Criteria:

* To have had a heart transplant, whenever
* To have an MRI scan of heart with measurement of T2 relaxation time (whatever the reason for examination)
* Major
* To be aware and cooperative
* Affiliation to social security plan
* To have given written consent after having received oral and written, clear and intelligible information

Exclusion Criteria:

* All contraindications to MRI (implantable defibrillator, cochlear implant, neurosurgical clip, intraorbital or encephalic metallic foreign body, endoprosthesis installed since less than 4 weeks, osteosynthesis materials installed since less than 6 weeks…)
* Instable hemodynamic status, acute respiratory failure, uncertain general status or necessity of continuous monitoring incompatible with MRI examination
* Minors or being under juridical protection or absence of social security
* Refusal or impossibility of informed consent of patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-08-31 (Actual); Primary Completion 2012-12-19 (Actual); Study Completion 2012-12-19 (Actual)

PRIMARY OUTCOMES:
Image quality assessed y senior radiologists | baseline
Movement correction in images assessed by senior radiologists | baseline

SECONDARY OUTCOMES:
Quantitative measurement of myocardial transversal relaxation time in 6 segments of short median axe cross-section of left ventricle in standard and ARTEMIS images | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No